CLINICAL TRIAL: NCT06755216
Title: Pelvis-Fetal Head Model With Applied Birth Simulation: Practical Training for Midwifery Students
Brief Title: Practical Birth Simulation for Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/1895; Individual Research Project. (Other: Karabük University)
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: MİDWİFERY STUDENT; Birth
Keywords: Midwifery; birth; model; raining

STUDY DESIGN:
Intervention Model Description: This is a two-group, parallel, prospective, and randomized controlled study.
Who Masked: Participant
Masking Description: Participants will not be aware of which group they have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): In order to identify students who meet the criteria for the study, the PIF and SSSCL will be administered as a pre-test to female students studying in the relevant departments of Karabük University Faculty of Health Sciences.
  After providing theoretical information to the students, the cardinal movements of the fetal head within the pelvis during the second stage of labor will be demonstrated in a laboratory setting. Students will be divided into groups of five, and after the demonstration, each student will be asked to perform all stages individually. Approximately 15 minutes will be allocated for each student. Two weeks later, the same students will be brought into the laboratory environment and asked to perform all procedural steps. While performing the steps, a researcher will mark the completed and missing actions on the learner's guide, and any missing steps will be explained to the student and corrected. For the post-test, the Learner's Guide (LG) and SSSCL will be administere
  Interventions: Behavioral: Experimantal group
- Control group (No Intervention): Students in both the control group will receive routine theoretical information. The cardinal movements of the fetal head within the pelvis during the second stage of labor will be explained. Afterwards, students will complete the pre-test using the personal information form (PIF) and Student Satisfaction and Self-Confidence Scale in Learning (SSSCL). Two weeks later, the students will be brought into the laboratory environment, where they will be asked to perform the practical steps of the theoretical lessons they have received, and a post-test will be administered. While performing the examination steps, a researcher will mark any omissions or completions on the learner's guide. In brief, students in the control group will receive regular theoretical information, and two weeks later, the examination steps and patient evaluation stages will be confirmed.

INTERVENTIONS:
Behavioral: Experimantal group — In order to identify students who meet the criteria for the study, the PIF and SSSCL will be administered as a pre-test to female students studying in the relevant departments of Karabük University Faculty of Health Sciences.
  After providing theoretical information to the students, the cardinal movements of the fetal head within the pelvis during the second stage of labor will be demonstrated in a laboratory setting. Students will be divided into groups of five, and after the demonstration, each student will be asked to perform all stages individually. Approximately 15 minutes will be allocated for each student. Two weeks later, the same students will be brought into the laboratory environment and asked to perform all procedural steps. While performing the steps, a researcher will mark the completed and missing actions on the learner's guide, and any missing steps will be explained to the student and corrected. For the post-test, the Learner's Guide (LG) and SSSCL will be administered
  Other Names: Intervention group
  Arms: Intervention group

SUMMARY:
Midwifery education consists of two parts: theoretical education and clinical training. Supporting clinical training is as important as theoretical training for the development of students' competencies. This simulation training, using the pelvis-fetal head model, will allow students to better understand the difficulties and complications they may encounter during childbirth and to develop the skills to intervene in these situations. This research is a pre-test post-test measurement, observational, randomized controlled study. The population of the research will consist of 3rd and 4th year students studying in the Midwifery department of Karabuk University Faculty of Health Sciences. The research sample will consist of 64 students studying in the 3rd and 4th year of midwifery. Work data will be collected using the Personal Information Form (PIF), Learner's Guide (LG), and Student Satisfaction and Self-Confidence Scale in Learning (SSSCL). Students in the control and experimental groups will be provided with routine theoretical knowledge. During the 2nd stage of labor, cardinal movements performed by the fetal head inside the pelvis will be explained. Subsequently, students will be asked to fill out the PIF and SSSCL for pre-testing. Two weeks later, students will be taken to the laboratory environment to perform the application steps for the theoretical lesson they received and a final test will be administered. While students carry out the examination steps, full-incomplete actions in the Learner's Guide will be marked by a researcher. In short, students in the control group will receive normal theoretical knowledge, and two weeks later, the examination steps and patient evaluation stages will be confirmed. The Study Group; After providing theoretical knowledge to the students, cardinal movements performed by the fetal head in the pelvis during the 2nd stage of labor will be explained practically in a laboratory environment. Students will be taken in groups of 5 and after the explanation of the application, each student will be asked to perform all stages individually. Approximately 15 minutes will be allocated for each student. Two weeks later, the same students will be taken to the laboratory and asked to perform all procedural steps. While students perform the procedural steps, any complete or incomplete applications will be marked by the researcher and then the incomplete applications will be explained to the student for them to complete. LG and SSSCL will be filled out for the final test. SPSS 27 package program will be used for data analysis, and a statistical significance level of 0.05 will be accepted for all analyses

DETAILED DESCRIPTION:
The second stage of labor involves cardinal movements of the fetal head within the pelvis. These movements ensure the head's alignment with the pelvis, facilitating rotation and easing delivery. It is important for midwifery students to learn these movements, as intervention may be necessary in case of any complications. Cardinal movements consist of seven key movements, and through these movements, the fetus navigates through the pelvis. Before interacting with pregnant women in clinical settings, it is crucial for midwifery students to master these cardinal and pelvic movements on a model. This ensures that, when in clinics and interacting with pregnant women, students can respond competently, confidently, and effectively. A study conducted by Tarrahi et al. (2022) found that simulation training can impact the performance of students, midwives, and gynecology residents. The increasing use of such training is also believed to improve safety for the pregnant woman, the postpartum mother, and the newborn, enhancing reliability.

This study is designed to reinforce the theoretical knowledge acquired by midwifery students, develop their practical skills, and foster competence through repeated opportunities for trial and error.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd or 4th-year Midwifery student, being between the ages of 18 and 25, voluntarily agreeing to participate in the study.

Exclusion Criteria:

* The ability to withdraw from the study at any time, being of male gender.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 65 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Student Satisfaction and Self-Confidence Scale in Learning (SSSCL) | 2 weeks
  This scale, published by the National League for Nurses (NLN), is used to measure students' attitudes and beliefs regarding simulation. The scale consists of two sub-dimensions, "satisfaction with learning" and "self-confidence," with a total of 13 items. The satisfaction with learning sub-dimension includes 5 items and measures satisfaction with the teaching method, diversity of learning materials, facilitation, motivation, and the overall appropriateness of the simulation. The self-confidence sub-dimension consists of 8 items and evaluates confidence in content sufficiency, content necessity, skill development, the availability of existing resources, and knowledge on how to seek help to solve clinical problems in the simulation. The 13th item of the scale is reverse scored.
  The response options for the scale are: 5 = Strongly agree, 4 = Agree, 3 = Neutral: Neither agree nor disagree, 2 = Disagree, 1 = Strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Yağmur Mutlu, Msc, Principal Investigator — Karabük University
Locations (1):
- Karabuk University, Karabük, Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided